CLINICAL TRIAL: NCT04146168
Title: Clinical and Patient-Centered Outcomes Three Years After Venaseal Treatment: Lake Washington Vascular VenaSeal Post Market Evaluation
Brief Title: Lake Washington Vascular VenaSeal™ Post-Market Evaluation
Acronym: New-WAVES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lake Washington Vascular (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-02
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Varicose Veins; Venous Reflux
Keywords: Venaseal; cyanoacrylate closure
MeSH Terms: conditions — Varicose Veins | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VenaSeal: Complete closure of previously treated veins will be assessed via ultrasound
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Closure of previously treated veins (with Venaseal) will be assessed via ultrasound.
  Other Names: Unilateral ultrasound of Limb

SUMMARY:
New-WAVES Study seeks to expand understanding/results from prior study (NCT02585726). Assessing both clinical outcomes and patient satisfaction after treatment with Venaseal/Cyanoacrylate Adhesive Closure System

DETAILED DESCRIPTION:
New WAVES is an investigator initiated protocol that will assess clinical outcomes and patient satisfaction after treatment with VenaSeal(TM)/ Cyanoacrylate Adhesive Closure System 3 years post-treatment. All patients treated from a multi-provider practice, whom meet protocol inclusion criteria, will be invited to consider participation in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years; 2. Treatment of the great, small or accessory saphenous vein or any combination of saphenous veins with the Venaseal Closure System; 3. Treatment occurred at least 30 months prior to study; 4. Ability to understand the requirements of the study and to provide informed consent.

-

Exclusion Criteria:

1. Subsequent treatment (such as laser or radiofrequency ablation) of venous disease in targeted vein segment after Venaseal closure; 2. Patients in whom index procedure information is unavailable; 3. Patients unwilling to undergo ultrasound evaluation and clinical examination of the previously treated limb; 4. Limbs that were treated in the VeClose trial (patients who participated in VeClose and later had contralateral limb treatment will be included).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the practice by identification of all patients treated with the Venaseal Closure System from October 2015 to December 31, 2016. This will include 50 prior subjects whom participated in the WAVES trial (ClinicalTrials.gov Identifier: NCT02585726), and up to 75 additional subjects whom also received the treatment with Venaseal but were not enrolled in the WAVES trial. All potential subjects for this study will have received treatment at Lake Washington Vascular, PLLC. Prior WAVES trial subjects initially enrolled will be approached with an introductory letter to be sent via e-mail or physical address. The correspondence will be sent to all potential study subjects explaining the purpose of the study and inviting them to participate. This correspondence will be followed up with a phone contact from study personnel.
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Complete Closure of Target Vein(s) at 3 years after index treatment | 3 years post treatment
  Complete closure is defined as Doppler Ultrasound examination showing closure along entire treated target vein segment with no discrete segments of patency exceeding 5 cm.

SECONDARY OUTCOMES:
Venous disease severity assessed via Venous Clinical Severity Score | 3 years post treatment
  Assessed via the revised Venous Clinical Severity Score (rVCSS). The rVCSS is an Investigator assessment of the severity of venous reflux disease, assessing signs and symptoms such as pain, varicose veins, venous edema, skin pigmentation, induration, and inflammation.
Clinical Severity via Varicose Vein Questionnaire (AVVQ) | 3 years post treatment
  Assessed via Aberdeen Varicose Vein Questionnaire (AVVQ) is a disease specific 13 item questionnaire is used to assess the impact of varicose veins on the quality of life, such as pain caused by varicose veins, and the need to take pain medication.
Quality of Life and Patient Satisfaction of Treatment: EQ-5D Questionnaire | 3 years post treatment
  Assessed via EQ-5D Questionnaire. The EQ-5D is a short generic quality of life survey that is commonly used outside of the United States for health technology assessments. The "health state today" question provides an overall assessment along a 20 cm visual analog scale (VAS) with a range from 0 ("worst imaginable health state") to 100 ("best imaginable health state").
Need for adjunctive treatments | 3 years post treatment
  Either at the index procedure or at any point following the index procedure
Health care utilization | 3 years post treatment
  Via chart review and patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Gibson, MD, Principal Investigator — Lake Washington Vascular, PLLC
Locations (3):
- United States (3):
  - Lake Washington Vascular, Bellevue, Washington
  - Lake Washington Vascular, Issaquah, Washington
  - Lake Washington Vascular, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No